CLINICAL TRIAL: NCT06356844
Title: The Effect of Adding Oral Resolvins to Patients Undergoing Transforaminal Epidural Steroid Injection for Low Back Pain Treatment"
Brief Title: The Effect of Resolvins on the Resolve of Inflammatory Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Aylin Ceren Sanli, Asist Dr, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27.02.2023-E.142568
Record Dates: First submitted 2024-03-05; First posted 2024-04-10 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain; Inflammatory Response; Lumbar Disc Herniation
Keywords: Transforaminal Steroid İnjection; Resolvin Therapy; Magnetic resonance imaging; Lumbar disc herniation; Cytokines level
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated with resolvin (Active Comparator): Transforaminal steroid injection with ultrasound and resolvin therapy
  Interventions: Dietary Supplement: Resolvin supplement
- No resolvin treatment (No Intervention): Transforaminal steroid injection with ultrasound and no resolvin treatment

INTERVENTIONS:
Dietary Supplement: Resolvin supplement — Transforaminal steroid injection will be administered to patients who are being followed up due to inflammatory low back pain. Patients will receive resolvin supplements for 6 months postoperatively.
  Arms: Treated with resolvin

SUMMARY:
Brief Summary: Inflammatory back pain is a chronic condition localized in the axial spine and sacroiliac joints.1 It often accompanies mechanical issues like lumbar disc herniation. While non-surgical interventions such as medication, physiotherapy, and epidural steroid injections are typically the initial approach, surgical options may be considered if these prove ineffective.2 Resolvins, derived from omega-3 fatty acids, have shown promise in reducing inflammation and pain. They help to resolve inflammatory responses, promote tissue repair, and decrease disc size, potentially reducing the need for surgery.3,4 This clinical trial aims to evaluate the efficacy of adding oral resolvins to transforaminal epidural steroid injections for treating lumbar disc herniation (LDH) The control group (Group C: n=25) will receive epidural steroids, while the study group (Group R: n=25) will receive both oral omega-3 supplementation and epidural steroids on the same day. Additionally, the study group will continue taking oral omega-3 supplements for six months.

The primary outcome measure will be changes in protruded/extruded disc size assessed via MRI, with secondary outcomes including pain levels measured by the Numeric Rating Scale (NRS) and serum cytokine levels (IL-6, IL-17, IL-1 beta, TNF-alpha) over the study period.

Discussion: This trial anticipates that combining the anti-inflammatory properties of resolvins with epidural steroid injection will provide a beneficial treatment for patients suffering from inflammatory low back pain.

DETAILED DESCRIPTION:
In the general population, about 70% to 80% of adults experience low back pain at some point in their lives. In primary care, the point prevalence ranges from 16% to 55%, making low back pain the most common neuropathic pain.5 In this context, radiculopathy is a common type of neuropathic pain. Pain can arise not only from direct mechanical pressure, such as from a herniated disc or degenerated bone, but also from inflammation and its associated proinflammatory cytokines. Inflammatory mediators contributing to neuropathic pain include nucleus pulpous cells and sequestered macrophages.6,7 Cytokines, as regulatory proteins acting as pro-inflammatory biomarkers, modulate the inflammatory response of all immune system cells during instances of inflammation.8 Despite its high prevalence, the response to medical treatment, physical therapy, and epidural steroid injections varies widely. For years, the widely accepted explanation for this variability has been the complex mechanisms involved in pain transmission. However, in recent years, it has been increasingly recognized that the lack of resolution of neuroinflammatory cells and mediators may be the most significant factor contributing to the varying treatment responses observed in individuals.9 Resolvins are specialized compounds derived from DHA (docosahexaenoic acid) and omega-3 fatty acids. Prior research indicates that certain resolvin subtypes, particularly D and E, aid in pain reduction by facilitating inflammation resolution. These specialized compounds, known as SPMs (Specialized pro-resolving mediators), regulate immune cell functions, modulate cytokine levels, and promote tissue repair mechanisms. 9,10 The aim of this study is to evaluate the impact of orally administered resolvins, in conjunction with epidural steroid injection, over a period of 6 months, on pain intensity and cytokine release during the remission phase. These effects will be assessed using magnetic resonance imaging.

Materials and Methods This clinical trial will be a randomized, controlled trial conducted at Bezmialem Vakıf University Hospital. A total of 30 patients will be enrolled in the study at this hospital. The study has received approval from the Ethics Boards of Bezmialem Vakif University Hospital. Prior to participation, all study participants will provide written informed consent.

Inclusion criteria: Patients must be classified as ASA I-II-III, aged between 18-75, presenting to the Algology department with low back pain due to lumbar disc herniation, have a pain intensity of ≥4 on the 0-10 scale pain NRS for low back pain, and/or experience radiating pain from the lower extremities caused by LDH (MRI scan confirmed lumbar disc herniation in our hospital).

Exclusion Criteria: Patients with known allergies to the drugs to be used in treatment, infection near the puncture site, known clotting disorders, alcohol and drug use, those who have used fish oil before, disorder of consciousness, liver failure, renal failure, advanced cardiac failure, uncontrolled diabetes mellitus, morbid obesity (body mass index (BMI) > 35 kg/m²), female patients during pregnancy and breastfeeding, not approving the informed consent form.

30 patients scheduled for caudal epidural injection, transforaminal epidural steroid injection will be included. Patients will be randomly assigned to two groups (Group K: control group, Group R: patients treated with resolvin) using opaque sealed envelopes. The physician performing the procedure (AT) and collecting data (AB) will be blinded to the groups. In Group R, treatment with 700 mg resolvin (omega DHA) will commence on the day the procedural decision is made.

Intervention: After the patient is admitted to the ward on the morning of the procedure, they will undergo routine blood tests, including a hemogram, APTT, INR, CRP, and sedimentation test. Once the results are obtained, the patient will be sent for the operation. Upon arrival in the operating room, basic monitoring including ECG, non-invasive blood pressure, and pulse oximetry will be performed. The operating room will be standardized, and normothermia will be maintained. Patients will be positioned prone on the operating table, and nasal oxygen support at 4L/min will be provided. After administering sedation and analgesia, prophylactic antibiotics will be given. The operative site will be prepared with an antiseptic solution and draped sterilely. All procedures are performed with the assistance of ultrasonography using a convex probe. After local anesthesia is applied to the areas to be treated, the procedure begins with a caudal epidural injection consisting of 40mg depomedrol, 60mg lidocaine, 20mg bupivacaine, and 100mg magnesium. Following this, the transforaminal epidural injection is administered with 2mg dexamethasone, 20mg lidocaine, 5mg bupivacaine, and 100mg magnesium. The same doses are applied to the facet insertion as the needle is withdrawn." After completion of the procedure, patients will be monitored in the recovery room for half an hour, followed by mobilization and transfer to the ward. Stable hemodynamics and absence of neurological deficits and any other complications (nausea, bradycardia, hypotension, urinary incontinence, drowsiness, bleeding, neurological deficit, edema, dyspeptic complaints due to fish oil or steroids) will warrant discharge after 6 hours.

Blood samples will be collected from the patients on the morning of the procedure day, during the one-week follow-up appointment after the procedure, and during the six-month follow-up along with MRI. Additionally, all medications used by patients during this period will be recorded.

Primary The primary objective of this study: Magnetic Resonance Imaging (MRI) is the gold standard for diagnosing lumbar disc herniation, with a diagnostic accuracy rate of 97%. It is also a crucial parameter used to determine the need for surgical intervention. MRI imaging will be used to measure the size of herniation preoperatively and at the 6th postoperative month by a radiologist who is blinded to the patient groups (AA).

Secondary objective of this study:

1. NRS Score: The Numeric Rating Scale (NRS) is a unidimensional scale using 11 numbers (ranging from 0 to 10) to assess pain intensity. Patients are asked to select the number that best represents their pain intensity, with 0 indicating no pain and 10 indicating the worst (unbearable) pain. Pain intensity will be assessed by having patients choose the number that corresponds to their pain intensity. Pain levels of all patients at the 1st postoperative week, 1st month, and 6th month will be recorded based on the NRS score by an anesthesiologist who is blinded to the patient groups.
2. Cytokines: Cytokines are small proteins synthesized by cells responsible for intercellular communication and interaction. They include various subtypes such as interleukins. The majority of studies found a positive association between the pro-inflammatory biomarkers CRP, IL-6, TNF-a, and low back pain. Blood tests for cytokine levels (Interleukin-6, Interleukin-17, Interleukin-1beta, TNF-alpha) were conducted preoperatively, at the 1st postoperative week, and at the 6th month by a medical biochemist who was blinded to the patient groups."

Statistics: Power analysis: Based on previous studies and considering an average difference of 0.50 units between groups with 80% power at a 95% confidence level, the minimum sample size was determined as 13 individuals per group, totaling 26 participants. Qualitative variables will be presented as numbers and percentages, while quantitative variables will be expressed as mean, standard deviation, median, minimum, and maximum. The relationships between qualitative variables will be examined using Pearson chi-square or Fisher exact chi-square tests. Normal distribution of quantitative variables will be assessed using the Kolmogorov-Smirnov test, and homogeneity of variance will be evaluated using the Levene test. Differences between the means of two independent groups will be analyzed using the Student's t-test, while median comparisons will be conducted using the Mann-Whitney U test. Paired t-tests and Wilcoxon signed-rank tests will be employed for comparing means and medians of two dependent groups, respectively. Following univariate analyses, appropriate regression analyses will be utilized based on the data structure. Calculations will be performed using the SPSS software package (version), with a statistical significance level set at 0.05.

Discussion: This trial anticipates that combining the anti-inflammatory properties of resolvins with epidural steroid injection will provide a beneficial treatment for patients suffering from inflammatory low back pain. This study demonstrates that two separate mechanisms result, including the decrease in cell recruitment to the inflammation site with steroids, which reflects an anti-inflammatory effect, and increases in cell exit with resolvin, which reflects a pro-resolution effect.

References

1. Lassiter W, Allam AE. Inflammatory Back Pain. Stat Pearls [Internet]. Treasure Island (FL): Stat Pearls Publishing; 2023 Jan-. 2022 Sep 5. PMID: 30969575.
2. Taso M, Sommernes JH, Kolstad F, Sundseth J, Bjorland S, Pripp AH, Zwart JA, Brox JI. A randomized controlled trial comparing the effectiveness of surgical and nonsurgical treatment for cervical radiculopathy. BMC Musculoskeletal Disorder. 2020 Mar 16;21(1):171. PMID: 32178655; PMCID: PMC7076994.
3. Ji RR, Xu ZZ, Strichartz G, Serhan CN. Emerging roles of resolvins in the resolution of inflammation and pain. Trends Neurosci. 2011 Nov;34(11):599-609. PMID: 21963090; PMCID: PMC3200462.
4. Liu C, Fan D, Lei Q, Lu A, He X. Roles of Resolvins in Chronic Inflammatory Response. Int J Mol Sci. 2022 Nov 28;23(23):14883. PMID: 36499209; PMCID: PMC9738788.
5. Yoshiaki Ota, Michael Connolly, Ashok Srinivasan, John Kim, Aristides A Capizzano, Toshio Moritani. Mechanisms and origins of spinal pain: from molecules to anatomy, with diagnostic clues and imaging findings Radiographic. Jul-Aug 2020;40(4):1163-1181.
6. Sowa GA, Coelho JP, Vo NV, Pacek C, Westrick E, Kang JD. Cells from degenerative intervertebral discs demonstrate unfavorable responses to mechanical and inflammatory stimuli: a pilot study. Am J Phys Med Rehabil 2012;91:846-855.
7. Videman T, Saarela J, Kaprio J, et al. Associations of 25 structural, degradative, and inflammatory candidate genes with lumbar disc desiccation, bulging, and height narrowing. Arthritis Rheum 2009;60:470-481.8
8. R van den Berg 1, E M Jongbloed 2, E I T de Schepper 2, S M A Bierma-Zeinstra 3, B W Koes 2, P A J Luijsterburg. The association between pro-inflammatory biomarkers and nonspecific low back pain: a systematic review Spine J 2018 Nov;18(11):2140-215
9. Ru-Rong Ji1, Zhen-Zhong Xu1, Gary Strichartz1, and Charles N. Serhan2. Emerging Roles of Resolvins in the Resolution of Inflammation and Pain. Trends Neurosci. 2011 November; 34(11): 599-609. doi:10.1016/j.tins.2011.08.005.
10. Chang Liu 1,2, Dancai Fan 3 , Qian Lei 1,3, Aiping Lu 1,4,5,* and Xiaojuan He 3,*. Roles of Resolvins in Chronic Inflammatory Response. Int. J. Mol. Sci. 2022, 23, 14883. https://doi.org/10.3390/ijms232314883.
11. Simon C, Le Corroller T, Pauly V, Creze M, Champsaur P, Guenoun D. Intradiscal oxygen-ozone therapy for the treatment of symptomatic lumbar disc herniation: A preliminary study. J Neuroradiol. 2022 Mar;49(2):180-186. doi: 10.1016/j.neurad.2021.09.004. Epub 2021 Oct 8. PMID: 34634298.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III
* Patients who underwent caudal epidural injection, facet joint injection and transforaminal injection due to lumbar disc herniation

Exclusion Criteria:

* Patients with known allergies to the drugs to be used in treatment
* Infection near the puncture site
* Known clotting disorders
* Alcohol and drug use
* Those who have used fish oil before
* Disorder of consciousness
* Liver failure, renal failure, advanced cardiac failure
* Uncontrolled diabetes mellitus
* Morbid obesity (body mass index (BMI) > 35 kg m-2)
* Female patients during pregnancy and breastfeeding
* Not approving the informed consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
changes in protruded/extruded disc size | Preoperatif, postoperative 6th month
  measure will be changes in protruded/extruded disc size assessed via MRI

SECONDARY OUTCOMES:
Pain intensity score | Preoperative, postoperative 1st week, postoperative 1th month, postoperative 6th month
  Postoperative pain assessed using a numeric rating scale 0 to 10 (0 = unsatisfied; 10 =very satisfied) and VAS (visual analogue scale)
Cytokine markers | Preoperative, postoperative 1st week, postoperative 6th month
  Evaluating Interleukin-6, Interleukin-17, Interleukin-1 beta, TNF-alpha marker results

CONTACTS AND LOCATIONS:
Overall Officials: zübeyde özdemir, Study Chair — ethics committee chairman
Locations (2):
- Turkey (Türkiye) (2):
  - Aylin Ceren Şanlı, Istanbul
  - Aylin Ceren, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
yes